CLINICAL TRIAL: NCT07270146
Title: A Multicenter, Randomized, Double-blind, Positive Drug Controlled Clinical Trial on the Efficacy and Safety of Guilu Erxian Oral Liquid in the Treatment of Oligozoospermia and Asthenospermia With Syndrome of Shen (Kidney) Essence Deficiency
Brief Title: Effectiveness and Safety of Guilu Erxian Oral Liquid in the Treatment of Oligozoospermia and Asthenospermia With Syndrome of Shen (Kidney) Essence Deficiency
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: DongE E Jiao Coporation Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DEEJ-CTP-20220129
Record Dates: First submitted 2025-11-24; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Mild and Moderate Oligozoospermia Asthenospermia or Oligoasthenospermia and the Syndrome Differentiation Type is Shen (Kidney) Essence Deficiency
MeSH Terms: conditions — Lymphoma, Follicular

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guilu Erxian Oral Liquid (Experimental)
  Interventions: Drug: Guilu Erxian Oral Liquid
- Wuzi Yanzong oral liquid (Active Comparator)
  Interventions: Drug: Wuzi Yanzong oral liquid

INTERVENTIONS:
Drug: Guilu Erxian Oral Liquid — Guilu Erxian Oral Liquid+Wuzi Yanzong Oral Liquid Simulator
  Arms: Guilu Erxian Oral Liquid
Drug: Wuzi Yanzong oral liquid — Wuzi Yanzong oral liquid+Guilu Erxian oral liquid simulator
  Arms: Wuzi Yanzong oral liquid

SUMMARY:
The main function of Guilu Erxian Oral Liquid is to warm the shen (kindney) and replenish essence. It is used for chronic shen (kindney) deficiency, waist and knee weakness, spermatorrhea and impotence. The treatment of deficiency of kidney essence and asthenospermia is to invigorate the shen (kindney) and replenish the essence, nourish the shen (kindney) and assist the essence. The idea of combining traditional Chinese and western medicine is to move the yang and calm the yin, and traditional Chinese medicine is mainly to invigorate the shen (kindney) and replenish the essence. In order to better provide the basis for clinical medication and meet the treatment needs of oligozoospermia and asthenospermia, this trial is intended to evaluate the effectiveness and safety of Guilu Erxian oral liquid in treating oligozoospermia and asthenospermia with Syndrome of Shen (Kidney) Essence Deficiency subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Married men aged 22 to 40;
2. Meet the diagnostic criteria of male infertility;
3. Meet the diagnostic criteria for mild and moderate oligozoospermia, asthenospermia and oligoasthenospermia;
4. Meet the TCM syndrome differentiation standard of Shen (kidney) essence deficiency syndrome;
5. Sign the informed consent form voluntarily.

Exclusion Criteria:

1. Infertility due to chromosome abnormalities (such as Roche heterotopia, Y chromosome microdeletion, etc.);
2. Varicocele or cryptorchidism;
3. Diseases affecting semen quality such as orchitis, epididymitis, mycoplasma and chlamydia infection;
4. Anejaculation, retrograde ejaculation and other sexual dysfunction;
5. Severe liver and kidney dysfunction (alanine aminotransferase (ALT)>1.5 × ULN, aspartate aminotransferase (AST)>1.5 × ULN, blood urea nitrogen (BUN)>2 × ULN, Cr>1 × ULN), disease of cardiovascular and cerebrovascular system, disease of hematopoietic system;
6. Hypertension (systolic blood pressure > 160 mmHg and / or diastolic blood pressure > 100 mmHg) or diabetes (fasting blood glucose > 7mmol / L) with poor drug control;
7. Serious mental illness, accompanied by mental disorder or loss of self-care ability;
8. Those who are allergic to the test drug;
9. Those who have long term bad habits such as smoking and drinking, which may affect fertility, or those who cannot ban smoking and drinking during the test, the specific criteria are as follows:

   ①History of smoking: Those who have smoked more than 5 cigarettes per day in the past 6 months;

   ②History of drinking: in the past 6 months, the average daily consumption of alcohol exceeded the following standards: 570 ml of beer, 200 ml of wine or 60 ml of spirit, each containing about 20 g of alcohol;
10. Those who have been unable to take the test drug in the past or have intolerable adverse reactions;
11. Those who used drugs to improve or affect sperm concentration or motility 1 month before screening;
12. Those who have participated in other clinical trials within 3 months before screening;
13. According to the judgment of the investigator, there are other persons who are not suitable to participate in this clinical trial.

Ages: 22 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 360 (Actual)
Dates: Start 2022-10-08 (Actual); Primary Completion 2025-02-10 (Actual); Study Completion 2025-02-10 (Actual)

PRIMARY OUTCOMES:
Total number of anterograde motile sperm (TPMSC) | 4,8,12 weeks after medical treatment
  Total number of anterograde motile sperm (TPMSC), the change value from the baseline

SECONDARY OUTCOMES:
Semen routine parameters: sperm concentration (SC), total sperm count (SPE-C), percentage of sperm forward movement (PR,%), total sperm vitality (PR+NP,%) | 4,8,12 weeks after medical treatment
  Semen routine parameters: sperm concentration (SC), total sperm count (SPE-C), percentage of sperm forward movement (PR,%), total sperm vitality (PR+NP,%), changes from baseline
TCM syndrome score | 4,8,12 weeks after medical treatment
  TCM syndrome score: the change value from the baseline
Pregnancy rate of spouse/partner | 4,8,12,24 weeks after medical treatment
  Pregnancy rate of the subject's spouse/partner
Male reproductive endocrine hormones: testosterone (T), follicle stimulating hormone (FSH), luteinizing hormone (LH), prolactin (PRL) | 12 weeks after medical treatment
  Male reproductive endocrine hormones: testosterone (T), follicle stimulating hormone (FSH), luteinizing hormone (LH), prolactin (PRL), the change value compared with the baseline (when it is conditional and necessary to conduct male reproductive endocrine hormone testing)
Sperm DNA fragment index, which is used for sperm DNA integrity analysis | 12 weeks after medical treatment
  Sperm DNA fragment index, which is used for sperm DNA integrity analysis, the change value compared with the baseline (when DFI detection is conditional and necessary)

CONTACTS AND LOCATIONS:
Locations (1):
- Xi Yuan Hospital of China Academy of Chinese Medical Sciences, Beijing, China